CLINICAL TRIAL: NCT05652023
Title: Noninvasive Ultrasound Assessment of Detrusor Dysfunction
Acronym: NUADD
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Azra Alizad, Principle Investigator, Mayo Clinic
Other Study IDs: 21-011734
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Bladder Dysfunction; Overactive Bladder; BPH With Urinary Obstruction
Keywords: Detrusor Pressure; Bladder Compliance; Ultrasound; Ultrasound Vibrometery
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to test a new ultrasound method called Quantitative Ultrasound Bladder Vibrometry to detect abnormal bladder function.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of quantitative ultrasound bladder vibrometry (QUBV) as a noninvasive tool for detrusor overactivity assessment and for benign prostatic hyperplasia (BPH) treatment selection. Participants in this study will have a QUBV ultrasound performed at the same time as a urodynamic study that had been ordered as part of their regular clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Aim1:

Age >18 scheduled to undergo UDS for their clinical care for one of the included diagnoses.

-Aim2: Inclusions: Age >45 scheduled to undergo selective photovaporization of the prostate.

Exclusion Criteria:

* Aim1:Obesity (BMI >35kg/m2), known neurologic disease impacting bladder function (e.g. spinal cord injury, multiple sclerosis, Parkinson's, prior cerebrovascular accident), previous pelvic radiation therapy, previous radical pelvic surgery (such as for uterine or colorectal cancer), prior bladder surgery (including prostate resection), and pregnant or breast-feeding women.
* Aim2:Obesity (BMI >35kg/m2), known neurologic disease impacting bladder function (e.g. spinal cord injury, multiple sclerosis, Parkinson's, prior cerebrovascular accident), previous pelvic radiation therapy, previous radical pelvic surgery (such as colorectal cancer).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aim 1:Cohort: Adults (male and female) with non-neurogenic lower urinary tract symptoms from one of the following conditions/symptoms: overactive bladder, benign prostatic hyperplasia, urinary frequency, incomplete bladder emptying, decreased force of urinary stream. N=200 Aim2:Cohort: Male adults with non-neurogenic lower urinary tract symptoms secondary to benign prostatic
Sampling Method: Probability Sample
Enrollment: 2023 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Accuracy of quantitative ultrasound vibrometry for measuring detrusor pressure | time Frame: Up to study completion, an average of 1 year
  Will be reported including 95% confidence intervals derived from the cross-validation procedure.

SECONDARY OUTCOMES:
Accuracy of quantitative ultrasound vibrometry for selecting BPH patients for de-obstructive surgery | time Frame: Up to study completion, an average of 1 year
  Will be reported including 95% confidence intervals derived from the cross-validation

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No